CLINICAL TRIAL: NCT03903211
Title: Longitudinal Changes of [18F]PI-2620 Positron Emission Tomography in Subjectives With Cognitively Normal, Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Longitudinal Changes of [18F]PI-2620 Positron Emission Tomography in Subjects With Cognitively Normal, Mild Cognitive Impairment and Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jae Seung Kim (Other)
Responsible Party: Sponsor-Investigator, Jae Seung Kim, Principal Investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI-18002
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Cognitively Normal; Mild Cognitive Impairment; Alzheimer Disease
Keywords: [18F]PI-2620; tauopathy; positron emission computed tomography
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Tauopathies | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitively normal individuals (Experimental): Cognitively normal individualswill receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620
- Subjects with Mild Cognitive Impairment (Experimental): Subjects with Mild Cognitive Impairment will receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620
- Subjects with Alzheimer Disease (Experimental): Alzheimer Disease Subjects with Alzheimer Disease will receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620

INTERVENTIONS:
Drug: [18F]PI-2620 — Imaging for evaluating the accumulation of abnormal tau protein in the brain
  Other Names: FluoroTau

SUMMARY:
The overall goal of this imaging trial is to evaluate crosssectional difference and longitudinal changes of [18F]PI-2620, a tau targeted positron emission computed tomography radioligand, in cognitively normal individuals, and subjects with mild cognitive impairment and Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. General Subject Inclusion Criteria

   In order to be eligible for participation in this trial, the subject must:
   * Be ≥ 40 and < 85 years of age at the Screening Visit.
   * Be able to read at a 6th grade level or equivalent, (as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation.)
   * Be able to speak, read, hear, and understand the language of the trial staff, and the informed consent form, and possess the ability to respond verbally to questions, follow instructions, and complete questionnaires and detailed neuropsychological test.
   * Have results of clinical laboratory tests/physical examination, vital signs, and ECG within normal limits (at 90 days prior to [18F]PI-2620 positron emission computed tomography) or clinically acceptable to the investigator at screening.
   * If female, not be of childbearing potential as indicated by one of the following
   * Each subject (or legal representative) must sign the informed consent form in accordance with local requirements after the scope and nature of the investigation have been explained to them, and before screening assessments.
2. Cognitively normal individuals
3. Subjects with Mild Cognitive Impairment
4. Subjects with Alzheimer Disease

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject fulfil any single criteria described below:

1. General Exclusion Criteria

   * Based on the investigators' judgement, if the patient is not capable of communicating with the site personnel, if the patient is not proficient in the language in which the psychometric tests will be completed, or if the patient is not sufficient for compliance with the study procedures.
   * The patient has an abnormal physical examination or abnormal laboratory test results at the screening that are clinically significant to affect results of the research, as judged by the investigator.
   * If the patient has or is suspicious of having a hypersensitivity or allergy to [18F] PI-2620 or its derivatives.
   * The patient is pregnant, is attempting to become pregnant, or is nursing (breast-feeding) children.
   * The patient has a history of alcoholism or drug dependency/abuse within the last 2 years before screening.
   * The patient has contraindications to undergo positron emission computed tomography or MRI, which include but are not restricted to the examples below: claustrophobia, cardiac pacemaker, metal devices around the eye or spinal cord, cochlear implant, etc.) at the screening visit.
   * The patient has been treated with any investigational medicinal product (IMP) within 1 years prior to the screening visit.
2. Cognitively normal individuals
3. Subjects with Mild Cognitive Impairment
4. Subjects with Alzheimer Disease

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Cross-sectional PI-2620 uptake measured by standard uptake value ratio (SUVR) | 60-90 minutes post injection
  Cross-sectional PI-2620 uptake measured by standard uptake value ratio (SUVR) in Cognitively normal, Mild Cognitive Impairment and Alzheimer Disease.

SECONDARY OUTCOMES:
Changes of PI-2620 uptake over time measured by standard uptake value ratios (SUVR) | 60-90 minutes post injection
  Changes of PI-2620 uptake over time measured by standard uptake value ratios (SUVR) in Cognitively normal, Mild Cognitive Impairment and Alzheimer Disease.
Correlation between standard uptake value ratio (SUVR) of [18F]PI-2620 positron emission computed tomography and neuropsychiatric test scores | 60-90 minutes post-injectio
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]PI-2620 positron emission computed tomography and scores of neuropsychiatric test
Correlation between standard uptake value ratio (SUVR) of [18F]PI-2620 positron emission computed tomography and indices of structural MRI | 60-90 minutes post injection
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]PI-2620 positron emission computed tomography and indices of structural Magnetic Resonance Imaging including cortical volume, hippocampal atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: JAE SEUNG KIM, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided